CLINICAL TRIAL: NCT02090686
Title: Efficacy of Pulsatile Cupping in Patients With Chronic Low Back Pain - a Randomized Controlled Study.
Brief Title: Pulsatile Cupping in Low Back Pain
Acronym: Cupping-LBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: HeVaTech GmbH (Unknown)
Responsible Party: Principal Investigator, Benno Brinkhaus, Prof., Charite University, Berlin, Germany
Allocation: Randomized | Masking: Single | Purpose: Treatment
Other Study IDs: Cupping-LBP
Record Dates: First submitted 2014-03-17; First posted 2014-03-18 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Pulsatile Cupping (Active Comparator)
  Interventions: Device: Pulsatile Cupping
- Minimal Cupping (Active Comparator)
  Interventions: Device: Minimal Cupping
- No Intervention (No Intervention): Waiting list

INTERVENTIONS:
Device: Pulsatile Cupping — 8 cupping sessions (each 8 minutes) in 4 weeks (-150 to -350 mbar), interval 2 seconds.
  Paracetamol on demand as rescue medication (maximum dosage 4 x500 mg/day)
  Other Names: HeVaTech PST 30 pulsatile cupping device
  Arms: Pulsatile Cupping
Device: Minimal Cupping — 8 cupping sessions (each 8 minutes) in 4 weeks witth (-60 to -70 mbar). Paracetamol on demand as rescue medication (maximum dosage 4 x500 mg/day).
  Other Names: HeVaTech PST 30 pulsatile cupping device
  Arms: Minimal Cupping

SUMMARY:
The purpose of this study is to determine whether pulsatile cupping with a cupping device is effective in the treatment of patients with chronic low back pain compared to no cupping or to minimal cupping.

ELIGIBILITY:
Inclusion Criteria:

* Male and female, 18-65 years
* Chronic low back pain (disease duration > 3 months)
* Pain intensity on visual analogue scale at inclusion > 40 mm (0-100 mm scale)
* Only pharmacological treatment with NSAID or no treatment in the last 4 weeks
* Undersigned informed consent form

Exclusion Criteria:

* Use of anticoagulants (Phenprocoumon, Heparin)
* Coagulopathy
* Cupping in the last 6 weeks
* Other CAM therapies in the last 12 weeks (e.g. acupuncture)
* Physical therapy in the last 12 weeks (e.g. massage, osteopathy)
* participation in another study in the last 3 months
* Paracetamol allergy or intolerance
* Pathological neurological symptoms such as muscular paralysis or paraesthesia due to spinal disc herniation or other causes
* Known renal and / or hepatic diseases
* Intake of central nervous system-acting analgesics in the last 6 weeks
* Applying for early retirement due to low back pain
* Severe disease that does not allow participation
* No undersigned informed consent form

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-03; Primary Completion 2014-10 (Actual); Study Completion 2015-02-28 (Actual)

PRIMARY OUTCOMES:
Intensity of pain on visual analogues scale | 4 weeks

SECONDARY OUTCOMES:
Intensity of pain on visual analogue scale | 12 weeks
Back function - FFbH-R-Questionnaire | 4 weeks, 12 weeks
Quality of Life - SF 36 | 4 weeks, 12 weeks
Assessment of perceived effect on Likert Scale | 4 weeks, 12 weeks
Intake of paracetamol | 4 weeks
Adverse events | week 1- 12

CONTACTS AND LOCATIONS:
Overall Officials: Benno Brinkhaus, Professor, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité Universitätsmedizin Berlin, Berlin, Germany

REFERENCES:
- [Derived] Teut M, Ullmann A, Ortiz M, Rotter G, Binting S, Cree M, Lotz F, Roll S, Brinkhaus B. Pulsatile dry cupping in chronic low back pain - a randomized three-armed controlled clinical trial. BMC Complement Altern Med. 2018 Apr 2;18(1):115. doi: 10.1186/s12906-018-2187-8. PMID 29609566